CLINICAL TRIAL: NCT03978169
Title: Pulmonary Impacts of Anaesthetic Modalities Evaluated by Ultrasound: A Prospective Study in Scheduled Knee Arthroplasty
Brief Title: Pulmonary Impacts of Anaesthetic Modalities Evaluated by Ultrasound
Acronym: PULCHO-KNEE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/18/0379
Record Dates: First submitted 2019-05-28; First posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Anesthesia
Keywords: anaesthetic modality; Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- General anaesthesia with orotracheal intubation: surgery patients under general anaesthesia with orotracheal intubation
  Interventions: Diagnostic Test: pleuropulmonary ultrasound
- General anaesthesia with laryngeal mask: surgery patient under general anaesthesia with laryngeal mask
  Interventions: Diagnostic Test: pleuropulmonary ultrasound
- Spinal anaesthesia: surgery's patients under Spinal anaesthesia
  Interventions: Diagnostic Test: pleuropulmonary ultrasound

INTERVENTIONS:
Diagnostic Test: pleuropulmonary ultrasound — three pleuro-pulmonary ultrasound scans will be performed, preoperatively on the day of surgery, post-operatively in the recovery room and the day after surgery

SUMMARY:
A prospective, observational, monocentric study aimed at identifying ultrasound changes in anaesthesia on the pulmonary parenchyma after knee arthroplastic surgery using the LUS score in the preoperative, immediate post-operative (D0) and late post-operative (D1) periods.

DETAILED DESCRIPTION:
Post-operative pulmonary complications are responsible from morbidity and mortality close to cardiovascular complications.

Perioperative and post-operative respiratory changes are secondary to anaesthesia (general anaesthesia, elongated position, tidal volume) and to surgery in particular abdominal and cardiothoracic surgery.

Several risk factors related to patients were identified: age, ASA score> 2, functional dependence, chronic obstructive pulmonary disease, congestive heart failure, obesity, smoking.

Pulmonary ultrasound is a simple and rapid means of monitoring, widely used in resuscitation and developing in anaesthesia.

The hypothesis of the study is that anaesthesia and / or ventilation is responsible for lung lesions observable by ultrasound from the recovery room, even after extra-thoracic surgeries.

To do this, it will perform 3 pleuro-pulmonary ultrasound scans, preoperatively on the day of surgery, post-operatively in the recovery room and the day after surgery. LUS score will be calculated. Preoperative data (morphology, comorbidities), preoperative (ventilation, filling, position, type of anaesthesia - general anaesthesia with intubation or laryngeal mask, spinal anaesthesia- , type of surgery) and postoperative data (constants, oxygen therapy, complications) will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing scheduled primary knee arthroplasty :
* Partial knee replacement surgery
* Total knee replacement surgery

  • Type of Anaesthesia
* General anaesthesia with orotracheal intubation
* General anaesthesia with laryngeal mask
* Spinal anaesthesia

  * Major Patient
  * Oral non opposition collected after oral information of the study

Exclusion Criteria:

* Refusal to participate
* Preoperative pleural pathology (pleural effusion, pleural symphysis)
* Pregnancy
* Patient under authorship or curators
* non-affiliation to a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergoing scheduled primary knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 99 (Estimated)
Dates: Start 2018-12-13 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
lung lesions by the anaesthetic and operative management after knee replacement surgery | 10 minutes before surgery
  Describe lung lesions by the anaesthetic and operative management after knee replacement surgery
lung lesions by the anaesthetic and operative management after knee replacement surgery | 10 minutes post surgery
  Describe lung lesions by the anaesthetic and operative management after knee replacement surgery
lung lesions by the anaesthetic and operative management after knee replacement surgery | 24hours post surgery
  Describe lung lesions by the anaesthetic and operative management after knee replacement surgery

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice FERRE, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- UHToulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided